CLINICAL TRIAL: NCT00723489
Title: A Study of the Systemic and Cutaneous Immune Responses to Yellow Fever Vaccination in Atopic Dermatitis Subjects
Brief Title: Immune Response to Yellow Fever Vaccination in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DAIT ADVN YF08; HHSN266200400029C
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Atopic Dermatitis
Keywords: Yellow Fever Vaccine; Scarification Method; Atopic Dermatitis; IgG antibodies
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YFV-17D (Right Deltoid) (Experimental): Participants will be randomized within each atopic dermatitis (AD) severity subgroup or as non-atopic controls to either subcutaneous (SC) or transcutaneous (TC) vaccine administration. In this arm, participants will receive a standard vaccine dose (5.5x10^4 Plaque Forming Units) of YFV-17D administered subcutaneously in the right deltoid and placebo vaccination transcutaneously (then covered with a semi-occlusive dressing) in the left deltoid. The site pharmacist will maintain the blind and an unblinded (i.e., masked) site coordinator will administer assigned treatment: investigators, participants and assessors remain blinded to treatment assignments throughout the duration of the trial.
  Interventions: Biological: Live Yellow Fever Vaccine (YFV-17D); Drug: YFV-17D Placebo
- YFV-17D (Left Deltoid) (Experimental): Participants will be randomized within each atopic dermatitis (AD) severity subgroup or as non-atopic controls to either subcutaneous (SC) or transcutaneous (TC) vaccination. In this arm, participants will receive YFV-17D vaccination (1x10^3 Plaque Forming Units) by transcutaneous administration (then covered with a semi-occlusive dressing to optimize YFV-17D absorption) in the left deltoid and placebo by subcutaneous administration in the right deltoid. The site pharmacist will maintain the blind and an unblinded (i.e., masked) site coordinator will administered treatment: investigators, participants and assessors remain blinded to treatment assignments throughout the duration of the trial.
  Interventions: Biological: Live Yellow Fever Vaccine (YFV-17D); Drug: YFV-17D Placebo

INTERVENTIONS:
Biological: Live Yellow Fever Vaccine (YFV-17D)
Drug: YFV-17D Placebo

SUMMARY:
The main objective of the Atopic Dermatitis and Vaccinia Immunization Network (ADVN) is to reduce the risk of the fatal reaction, eczema vaccinatum (EV), to the smallpox vaccination in those with atopic dermatitis (AD). Since vaccination with live vaccinia virus (VV) in individuals with AD increases the risk of EV, a yellow fever vaccine was chosen. The purpose of this study is to determine the immune response to a yellow fever vaccine in adults with AD.

DETAILED DESCRIPTION:
AD is a chronic inflammatory skin disorder characterized by recurrent viral skin infections. The purpose of this study is to understand the immune response to a yellow fever vaccine in adults with AD. This study will provide substantial information about normal and defective cutaneous immunity in participants with AD in response to a live virus vaccine, which is critical for understanding the EV reaction.

An individual's participation in the study will last up to 13 weeks. Participants will be randomized into one of two arms. The first experimental arm will consist of 20 adults with AD and 20 healthy adults. They will receive one dose of YFV-17D by subcutaneous administration in the right deltoid and receive one dose of YFV-17D placebo by transcutaneous administration in the left deltoid. The second arm will consist of 20 adults with AD and 20 healthy adults. They will receive one dose of YFV-17D placebo by subcutaneous administration in the right deltoid and receive one dose of YFV-17D vaccine transcutaneously in the left deltoid.

This study will consist of 6 follow-up visits over a 35 day period after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Atopic Dermatitis or Non-atopic control
* Born and currently residing in the United States
* Weight of at least 110 lbs at the Screening Visit
* Not previously vaccinated for YFV, tick-borne encephalitis (TBEV), Japanese encephalitis virus (JEV), or dengue fever
* Agree to use adequate contraception 30 days prior to and until their participation in the study is completed. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* AD subjects with exfoliative erythroderma or lacking a minimum 10 cm diameter area of normal appearing skin on the deltoid or thigh vaccination sites
* Have a body mass index (BMI) of 30 or greater at the Screening Visit
* Known history of infection with YFV, dengue fever, TBEV, JEV, or West Nile Virus (WNV)
* A family history of severe reactions to the yellow fever vaccine
* Traveled to Africa or South America (including participants who plan to travel to these areas prior to completion of the study)
* History of egg allergy or have a positive egg allergy skin prick test that is administered at the Screening visit
* History of acute hypersensitivity reaction to any components of the yellow fever vaccine (including gelatin)
* Have latex allergy
* Have lidocaine allergy
* Are allergic or hypersensitive to TegadermTM
* Received systemic immunosuppressants within 30 days prior to receiving the vaccination
* Received systemic corticosteroids, anti inflammatory biologics (e.g., alefacept, etanercept, etc.), or calcineurin inhibitors within 30 days prior to receiving the vaccination
* Received systemic antibiotics or antivirals within 7 days of receiving the vaccination
* Received greater than 440 mcg of inhaled steroids per day within 6 months prior to receiving the vaccination
* Received Xolair (Omalizumab) within 1 year prior to receiving the vaccination
* Received immunotherapy within 30 days prior to receiving the vaccination
* Received any vaccine within 30 days prior to randomization or expected receipt 30 days after randomization
* Received topical antibiotics, antivirals, immune enhancers (e.g., imiquimod), or calcineurin inhibitors within 7 days prior to receiving the vaccination
* Received topical corticosteroids within 7 days prior to receiving the vaccination
* Received phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA]) within 30 days prior to receiving the vaccination
* Acute febrile illness or active fungal, bacterial, or viral infections (subjects may be reconsidered for enrollment once the condition has resolved)
* Skin disease other than AD that might compromise the stratum corneum barrier (e.g., clinically evident ichthyosis, bullous disease, psoriasis)
* Current or past history of malignancy or of autoimmune or immunodeficiency diseases. More information on this criterion can be found in the protocol.
* Pregnant or breastfeeding
* Have an anti-nuclear antibody (ANA) titer that is equal to or greater than 1/160 at the Screening Visit
* Have a serum immunoglobulin (Ig)G, IgM, IgA, C3, or C4 level below the normal range at the Screening Visit
* Have a manual lymphocyte count that is less than 1000 lymphocytes per microliter

Ages: 27 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Hanifin, M.D., Study Chair — Oregon Health and Science University; Mark Slifka, Ph.D., Principal Investigator — Oregon Health and Science University; Eric Simpson, M.D., Principal Investigator — Oregon Health and Science University; Henry Milgrom, M.D., Principal Investigator — National Jewish Health; Richard Gallo, M.D., Ph.D., Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Derived] Slifka MK, Leung DY, Hammarlund E, Raue HP, Simpson EL, Tofte S, Baig-Lewis S, David G, Lynn H, Woolson R, Hata T, Milgrom H, Hanifin J. Transcutaneous yellow fever vaccination of subjects with or without atopic dermatitis. J Allergy Clin Immunol. 2014 Feb;133(2):439-47. doi: 10.1016/j.jaci.2013.10.037. Epub 2013 Dec 10. PMID 24331381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 2008 to March 2011, three centers in the United States recruited participants ages 27 to 43 years who fulfilled eligibility criteria. Refer to the Eligibility Section for more details.
Groups:
- YFV-17D SC - (Non-AD): Healthy volunteer participants who did not have atopic dermatitis defined by Atopic Dermatitis and Vaccinia Network (ADVN) Standard Diagnostic Criteria and received a 0.5 mL dose of the Yellow Fever vaccine (YFV-17D) by subcutaneous (SC) administration in the right deltoid and one dose of placebo by transcutaneous (TC) administration in the left deltoid.
- YFV-17D SC - (AD): Participants classified as atopic dermatitis (AD) defined by the Atopic Dermatitis and Vaccinia Network (ADVN) Standard Diagnostic Criteria and received a 0.5 mL dose of YFV-17D by subcutaneous administration in the right deltoid and one dose of placebo by transcutaneous administration in the left deltoid.
- YFV-17D TC - (Non-AD): Healthy volunteer participants who did not have atopic dermatitis defined by the Atopic Dermatitis and Vaccinia Network (ADVN) Standard Diagnostic Criteria and received one dose of YFV-17D vaccine by transcutaneous administration in the left deltoid and one dose of placebo by subcutaneous administration in the right deltoid.
- YFV-17D TC - (AD): Participants classified as atopic dermatitis (AD) and defined by the Atopic Dermatitis and Vaccinia Network (ADVN) Standard Diagnostic Criteria received one dose of YFV-17D vaccine by transcutaneous administration in the left deltoid and one dose of placebo by subcutaneous administration in the right deltoid.
Period: Overall Study
Arm/Group | YFV-17D SC - (Non-AD) | YFV-17D SC - (AD) | YFV-17D TC - (Non-AD) | YFV-17D TC - (AD)
Started | 21 | 19 | 19 | 23
Completed | 20 (Includes seroconverters and non-seroconverters) | 15 (Includes seroconverters and non-seroconverters) | 19 (Includes seroconverters and non-seroconverters) | 20 (Includes seroconverters and non-seroconverters)
Not Completed | 1 | 4 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Seropositive at baseline | 1 | 0 | 0 | 0
Not completed — Prohibited Medication | 0 | 0 | 0 | 1
Not completed — Samples Collected Out of Window | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | YFV-17D SC - (Non-AD) | YFV-17D SC - (AD) | YFV-17D TC - (Non-AD) | YFV-17D TC - (AD) | Total
Number analyzed (Participants) | 20 | 15 | 19 | 20 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (4.5) | 34.7 (6.2) | 33.9 (4.7) | 32.8 (4.3) | 33.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 10 | 12 | 42
  Male | 8 | 7 | 9 | 8 | 32
Region of Enrollment [Number; unit: participants]
  United States | 20 | 15 | 19 | 20 | 74
Total Serum Immunoglobulin E (IgE; kU/L) [Mean (Standard Deviation); unit: kU/L] — Total amount of IgE in the blood, which is a measurement of allergen sensitization. Higher IgE is indicative of greater allergen sensitization. There is no "normal" level for total serum IgE since a wide overlap exists between the total serum IgE in healthy non-allergic and allergic individuals.
  kU/L | 35.4 (40.3) | 1166.4 (3609.5) | 73.6 (115.7) | 2742.1 (8262.5) | 1006.0 (4646.1)
Percent Eosinophils in Blood [Mean (Standard Deviation); unit: Percent Eosinophils] — Eosinophils are a type of immune cell that has granules (small particles) with enzymes that are released during infections, allergic reactions, and asthma. An eosinophil is a type of white blood cell. Normal Reference Range: 0.0% - 7.0%.
  Percent Eosinophils | 2.6 (1.9) | 3.7 (2.1) | 2.4 (2.0) | 3.8 (3.2) | 3.1 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Anti-YF Antibody Levels by Measurement of Log10 Neutralization Index (LNI): YFV-17D TC- (AD) Participants Compared to YFV-17D TC- (Non-AD) Participants
Description: Log10 Neutralization Index (LNI) is the Log10 difference in virus titer (measurement of amount of virus) between pre-vaccination and post-vaccination. An LNI greater than or equal to 0.7 suggests that a person has active immunity against Yellow Fever virus.
Time Frame: 30 days after Yellow Fever (YF) immunization (Acceptable Blood Draw Range: Day 28 - Day 35 after YF immunization)
Population: All participants who completed the study; and seroconverted
Measure: Mean (Standard Deviation); unit: LNI
Arm/Group | YFV-17D TC - (AD) | YFV-17D TC - (Non-AD)
Number analyzed (Participants) | 18 | 14
LNI | 1.8 (0.4) | 1.8 (0.4)
Statistical Analysis 1: Comparison: YFV-17D TC - (AD) vs YFV-17D TC - (Non-AD); Test type: Superiority or Other; p = 0.86, ANOVA — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.3 to 0.2] — Mean (AD) - Mean (Non-AD)

2. Primary Outcome: Comparison of Anti-YF Antibody Levels by Measurement of Log10 Neutralization Index (LNI): YFV-17D SC - (AD) Participants Compared to YFV-17D SC- (Non-AD) Participants
Description: as for outcome 1
Time Frame: 30 days after YF immunization (Acceptable Blood Draw Range: Day 28 - Day 35 after Yellow Fever immunization)
Population: All participants who completed the study; and seroconverted
Measure: Mean (Standard Deviation); unit: Log10 Neutralization Index (LNI)
Arm/Group | YFV-17D SC - (AD) | YFV-17D SC - (Non-AD)
Number analyzed (Participants) | 14 | 20
Log10 Neutralization Index (LNI) | 1.8 (0.3) | 1.8 (0.3)
Statistical Analysis 1: Comparison: YFV-17D SC - (AD) vs YFV-17D SC - (Non-AD); Test type: Superiority or Other; p = 0.86, ANOVA — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.2 to 0.2] — Mean (AD) - Mean (Non-AD)

3. Primary Outcome: Comparison of Anti-YF Antibody Levels by Measurement of Log10 Neutralizing Titer 50 (NT50): YFV-17D TC - (AD) Participants Compared to YFV-17D TC - (Non - AD) Participants
Description: Neutralization titer (NT50) is the dilution of serum (antibody) that results in a 50% reduction in the amount of virus. A higher NT50 number reflects the presence of more protective antibody levels against the Yellow Fever virus. Some studies have used an NT50 titer of 1:10 or 1:20 as the minimum level to suggest that a person has active immunity against the Yellow Fever virus.
Time Frame: 30 days after Yellow Fever (YF) immunization (Acceptable Blood Draw Range: Day 28 - Day 35 after YF immunization)
Population: All participants who completed the study; and seroconverted
Measure: Mean (Standard Deviation); unit: Log10 (NT50)
Arm/Group | YFV-17D TC - (AD) | YFV-17D TC - (Non-AD)
Number analyzed (Participants) | 18 | 14
Log10 (NT50) | 3.5 (0.4) | 3.8 (0.3)
Statistical Analysis 1: Comparison: YFV-17D TC - (AD) vs YFV-17D TC - (Non-AD); Test type: Superiority or Other; p = 0.10, ANOVA — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.05] — Mean (AD) - Mean (Non-AD)

4. Primary Outcome: Comparison of Anti-YF Antibody Levels by Measurement of Log10 Neutralizing Titer 50 (NT50): YFV-17D SC - (AD) Participants Compared to YFV-17D SC - (Non-AD) Participants
Description: as for outcome 3
Time Frame: 30 days after Yellow Fever (YF) immunization (Acceptable Blood Draw Range: Day 28 - Day 35 after YF immunization)
Population: All participants who completed the study; and seroconverted
Measure: Mean (Standard Deviation); unit: Log10 (NT50)
Arm/Group | YFV-17D SC - (AD) | YFV-17D SC - (Non-AD)
Number analyzed (Participants) | 14 | 20
Log10 (NT50) | 3.6 (0.4) | 3.5 (0.3)
Statistical Analysis 1: Comparison: YFV-17D SC - (AD) vs YFV-17D SC - (Non-AD); Test type: Superiority or Other; p = 0.66, ANOVA — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.3] — Mean (AD) - Mean (Non-AD)

5. Secondary Outcome: Comparison of Count of Seroconverters: YFV-17D TC- (AD) Participants Compared to YFV-17D TC - (Non-AD) Participants
Description: Seroconversion is defined as a Log10 Neutralization Index (LNI) of 0.7 or higher. A value greater than or equal to 0.7 suggests that a person has active immunity against Yellow Fever virus.
Time Frame: Day 0 to Day 30 (Acceptable Post-Vaccination Blood Draw Range: Day 28 - Day 35)
Population: Includes all participants who completed the study; seroconverters as well as non-seroconverters
Measure: Number; unit: participants
Arm/Group | YFV-17D TC - (AD) | YFV-17D TC - (Non-AD)
Number analyzed (Participants) | 20 | 19
participants
  Did not seroconvert | 2 | 5
  Seroconverted | 18 | 14
Statistical Analysis 1: Comparison: YFV-17D TC - (AD) vs YFV-17D TC - (Non-AD); Test type: Superiority or Other; p = 0.24, Fisher Exact — P-value is not adjusted for multiple comparisons

6. Secondary Outcome: Comparison of Count of Seroconverters: YFV-17D SC - (AD) Participants Compared to YFV-17D SC - (Non-AD) Participants
Description: as for outcome 5
Time Frame: Day 0 to Day 30 (Acceptable Post-Vaccination Blood Draw Range: Day 28 - Day 35)
Population: Includes all participants who completed the study; seroconverters as well as non-seroconverters
Measure: Number; unit: participants
Arm/Group | YFV-17D SC - (AD) | YFV-17D SC - (Non-AD)
Number analyzed (Participants) | 15 | 20
participants
  Did not seroconvert | 1 | 0
  Seroconverted | 14 | 20
Statistical Analysis 1: Comparison: YFV-17D SC - (AD) vs YFV-17D SC - (Non-AD); Test type: Superiority or Other; p = 0.43, Fisher Exact — P-value is not adjusted for multiple comparisons

7. Secondary Outcome: Comparison in Log10 Transformed Lymphocyte Count on Day 30 Post YF Immunization: IFN-gamma Positive, Tumor Necrosis Factor- Alpha (TNF Alpha) Positive, CD4 Positive T-cells, YFV-17D SC - (AD) Compared to YFV-17D SC - (Non- AD) Participants
Description: Comparison by designated reporting groups: the Log10 transformed lymphocyte count of CD4 Positive T-cells expressing IFN-gamma and TNF-alpha in every 10^6 CD4 Positive T-cells on Day 30 (acceptable blood draw window: Day 28 - 35).
Time Frame: Day 30 (Day 28-35)
Population: Analysis excludes 1 SC-(AD) participant who did not seroconvert, 1 SC-(Non-AD) participant whose samples were collected out of window, and 3 SC (Non-AD) and 1 SC-(AD) due to problems with sample processing
Measure: Mean (Standard Deviation); unit: Log10 cell count/10^6 cells
Arm/Group | YFV-17D SC - (AD) | YFV-17D SC - (Non-AD)
Number analyzed (Participants) | 13 | 16
Log10 cell count/10^6 cells | 2.8 (0.4) | 2.7 (0.3)
Statistical Analysis 1: Comparison: YFV-17D SC - (AD) vs YFV-17D SC - (Non-AD); This analysis excludes 1 SC-(AD) participant who did not seroconvert. Only participants who had peripheral blood T-cell samples collected from Day 0 to Day 30 as specified in the Outcome Measure Time Frame were included in analysis (1 SC -(Non-AD) participant was excluded). T-cell data from 3 SC-(Non-AD) and 1 SC-(AD) participant was excluded due to problems with sample processing; Test type: Superiority or Other; p = 0.48, Mixed Models Analysis — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) Day 30 = 0.1, 95% CI 2-sided [-0.1 to 0.3] — Mean (AD) - Mean (Non-AD)

8. Secondary Outcome: Comparison in Log10 Transformed Lymphocyte Count on Day 30 Post YF Immunization: IFN-gamma Positive, Tumor Necrosis Factor- Alpha (TNF Alpha) Positive , CD4 Positive T-cells, YFV-17D TC - (AD) Compared to YFV-17D TC - (Non-AD) Participants
Description: Comparison by designated reporting groups: the Log10 transformed count of CD4 Positive T-cells that express IFN-gamma and TNF-alpha in every 10^6 CD4 Positive T- Cells (Day 30). A higher count reflects a better immune response to Yellow Fever virus.
Time Frame: Day 30 (Day 28-35)
Population: Participants who did not seroconvert were excluded from this analysis (2 TC-(AD) and 5 TC-(Non-AD)). T-cell data from 4 TC-(AD) and 3 TC-(Non-AD) subjects was excluded due to problems with sample processing
Measure: Mean (Standard Deviation); unit: Log10 cell count/10^6 cells
Arm/Group | YFV-17D TC - (AD) | YFV-17D TC - (Non-AD)
Number analyzed (Participants) | 14 | 11
Log10 cell count/10^6 cells | 2.5 (0.3) | 2.7 (0.2)
Statistical Analysis 1: Comparison: YFV-17D TC - (AD) vs YFV-17D TC - (Non-AD); Participants who did not seroconvert were excluded from this analysis (2 TC-(AD) and 5 TC-(Non-AD)). T-cell data from 4 TC-(AD) and 3 TC-(Non-AD) subjects was excluded due to problems with sample processing; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) Day 30 = -0.3, 95% CI 2-sided [-0.5 to -0.02] — Mean (AD) - Mean (Non-AD)

9. Secondary Outcome: Comparison in Log10 Transformed Lymphocyte Count on Day 30 Post YF Immunization: IFN-gamma Positive, Tumor Necrosis Factor- Alpha (TNF Alpha) Positive, CD8 Positive T-cells, YFV-17D SC -(AD) Compared to YFV-17D SC - (Non-AD) Participants
Description: Comparison by designated reporting groups: the Log10 transformed lymphocyte count of CD8 Positive T-cells expressing IFN-gamma and TNF-alpha in every 10^6 CD8 Positive T-cells.
Time Frame: Day 30 (Day 28-35)
Population: Analysis excludes 1 SC-(AD) participant who did not seroconvert, 1 SC-(AD) participant whose samples were collected out of window, and 3 SC (Non-AD) and 1 SC-(AD) due to problems with sample processing
Measure: Mean (Standard Deviation); unit: Log10 cell count/10^6 cells
Arm/Group | YFV-17D SC - (AD) | YFV-17D SC - (Non-AD)
Number analyzed (Participants) | 13 | 16
Log10 cell count/10^6 cells | 3.4 (0.3) | 3.3 (0.4)
Statistical Analysis 1: Comparison: YFV-17D SC - (AD) vs YFV-17D SC - (Non-AD); [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) Day 30 = 0.04, 95% CI 2-sided [-0.3 to 0.4] — Mean (AD) - Mean (Non-AD)

10. Secondary Outcome: Comparison in Log10 Transformed Lymphocyte Count on Day 30 Post YF Immunization: IFN-gamma Positive, Tumor Necrosis Factor- Alpha (TNF Alpha) Positive, CD8 Positive T-cells, YFV-17D TC - (AD) Compared to YFV-17D TC - (Non-AD) Participants
Description: Comparison by designated reporting groups: the Log10 transformed count of CD8 Positive T-cells expressing IFN-gamma and TNF-alpha in every 10^6 CD8 Positive T-cells.
Time Frame: Day 30 (Day 28-35)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Log10 cell count/10^6 cells
Arm/Group | YFV-17D TC - (AD) | YFV-17D TC - (Non-AD)
Number analyzed (Participants) | 14 | 11
Log10 cell count/10^6 cells | 3.0 (0.5) | 3.3 (0.5)
Statistical Analysis 1: Comparison: YFV-17D TC - (AD) vs YFV-17D TC - (Non-AD); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis — P-value is not adjusted for multiple comparisons; Mean Difference (Final Values) Day 30 = -0.4, 95% CI 2-sided [-0.7 to -0.01] — Mean (AD) - Mean (Non-AD)

ADVERSE EVENTS:
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Arm/Group | YFV-17D SC - (Non-AD) | YFV-17D SC - (AD) | YFV-17D TC - (Non-AD) | YFV-17D TC - (AD)
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 20/21 | 19/19 | 18/19 | 21/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | YFV-17D SC - (Non-AD) (N=21) | YFV-17D SC - (AD) (N=19) | YFV-17D TC - (Non-AD) (N=19) | YFV-17D TC - (AD) (N=23)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Application site pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Fatigue (General disorders) | 3 (3) | 7 (9) | 0 (0) | 7 (8)
Injection site pain (General disorders) | 4 (4) | 2 (3) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Blood cholesterol increased (Investigations) | 4 (4) | 5 (6) | 4 (5) | 3 (3)
Blood glucose decreased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Blood glucose increased (Investigations) | 2 (2) | 1 (1) | 4 (5) | 5 (5)
Blood magnesium decreased (Investigations) | 5 (5) | 2 (3) | 9 (11) | 4 (5)
Haemoglobin decreased (Investigations) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Lymph node palpable (Investigations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2) | 4 (4) | 3 (3) | 5 (5)
Neutrophil count decreased (Investigations) | 9 (9) | 5 (5) | 5 (6) | 5 (5)
White blood cell count decreased (Investigations) | 2 (2) | 3 (3) | 4 (4) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 5 (6) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (4) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (11) | 4 (5) | 2 (2) | 6 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 5 (6) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No